CLINICAL TRIAL: NCT06427291
Title: A Phase I, Open Label, Multiple Dose, Dose Escalation and Expansion Study to Evaluate the Safety and Efficacy of T3011 in Patients With BCG-Failure Non-Muscle-Invasive Bladder Cancer (NMIBC)
Brief Title: Clinical Study of T3011 Intravesical Instillation for Treatment of NMIBC Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ding-Wei Ye, Principal Investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MVR-T3011-ES-EC61-UC
Record Dates: First submitted 2024-05-16; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Bladder Cancer
Keywords: high-risk non-muscle invasive bladder cancer (NMIBC); BCG failure or intolerance
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Herpes virus T3011 injection (Experimental): T3011 with the dose of 5 x 10^7 PFU, 5 x 10^8 PFU or 2 x 10^9 PFU is administered via intravesical instillation, once a week (QW) for the first 12 weeks and then every 2 weeks (Q2W) until 12 months.
  Interventions: Biological: Herpes virus T3011 injection

INTERVENTIONS:
Biological: Herpes virus T3011 injection — T3011 will be instilled in the entire solution volume of 50ml, and be will be left in the bladder for at least 1 hour, no more than 2 hours. After competing instillation, the patients should be instructed to drink at lest 1000mL of water

SUMMARY:
This is a prospective, open-label, single-arm investigator-initiated clinical study. It is used to evaluate the safety and efficacy of T3011 intravesical instillation in patients with BCG-failure high-risk non-muscle invasive bladder cancer (NMIBC)

ELIGIBILITY:
Inclusion Criteria:

1. Participants who understand and voluntarily sign the written ICF, and are willing and able to comply with all trial requirements.
2. Male or female, aged ≥ 18 years at the time of signing the ICF.
3. Participants with a histologically confirmed diagnosis of NMIBC (Ta, T1 and/or Tis).
4. Participants with high risk NMIBC who have been diagnosed by cystoscopy, urine cytology, and histopathology within 8 weeks prior to the first dose administration and have failed or intolerant to BCG treatment after TURBT surgery, and are not suitable or willing to undergo radical cystectomy.
5. BCG-failure include BCG refractory, recurrence or relapsing after BCG treatment, BCG unresponsive and BCG intolerant.
6. All tumors should have no visible tumors after transurethral bladder tumor resection (TURBT). If meeting the requirements for secondary resection, secondary resection need to be done. It is recommended to perform secondary resection if the following conditions are met: the first TURBT is insufficient, there is no muscle tissue in the first resection specimen (excluding low-grade [Ta G1] tumors and pure in situ cancers), T1 stage tumors, and high-grade [G3] tumors (excluding pure in situ cancers); Secondary resection is recommended to be performed 2-6 weeks after the first resection; Participants undergoing secondary resection must meet the requirement of no visible tumors after surgery.
7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1.
8. Expected survival ≥3 months.
9. Sufficient hematology and terminal organ function were met within 4 weeks prior to the first s treatment, for example, having sufficient bone marrow reserves and organ function:

   * Hematology (hematopoietic growth factor treatment or blood transfusion should not be given within 2 weeks prior to the treatment of study drug): ANC≥1.5×10^9/L, PLT count ≥75×10^9/L, Hemoglobin (HGB) ≥90 g/L.
   * Renal function: Creatinine clearance ≥60 mL/min (based on Cockcroft-Gault equation for calculation)
   * Hepatic function: Serum total bilirubin (TBIL) ≤1.5×ULN, Aspertate aminotransferase (AST) and alanine transaminase (ALT) ≤3×ULN
   * Coagulation function: International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN; Activated partial thromboplastin time (aPTT) ≤1.5×ULN
10. Women with fertility should agree to use contraceptive measures (such as intrauterine devices (IUDs), contraceptives, or condoms) during the study period and within 6 months after the end of the study; Within 7 days prior to enrollment in the study, the serum or urine pregnancy test was negative and must be a non lactating patient; Men should agree to patients who must use contraceptive measures during the study period and within 6 months after the end of the study period. Note: A female subject with fertility is defined as a female subject who has not reached a postmenopausal state after menarche (continuous amenorrhea for at least 12 months, with no other clear cause other than menopause), and has not undergone surgery (i.e. bilateral ovariectomy, fallopian tube resection, and/or hysterectomy) or other causes determined by the researcher (such as underdeveloped Mullerian tubes) leading to permanent infertility.

Exclusion Criteria:

Patients meeting one or more of the following criteria will be excluded:

1. The diagnosis is confirmed as muscle invasive bladder cancer (T2-T4).
2. Patients with concurrent upper and lower urinary tract epithelial carcinoma, lymph node metastasis, or distant metastasis.
3. Pregnant and lactating female patients.
4. Having major surgery within 4 weeks prior to the first dose of the study drug, or anticipate the need for major surgery rather than diagnosis after enrolling the study.
5. In addition to immediate instillation therapy after TURBT surgery, anti-tumor drug treatments such as chemotherapy, radiation therapy, biological therapy, endocrine therapy, targeted therapy, immunotherapy, etc. have been received within 4 weeks prior to the first dose of the study drug (excluding nitroso urea, mitomycin C, oral fluorouracil, small molecule targeted drugs, and traditional Chinese medicine with anti-tumor indications). Nitrso urea or mitomycin C is within 6 weeks prior to the first use of the study drug, and oral fluorouracil and small molecule targeted drugs are within 2 weeks prior to the first use of the study drug or within 5 half-lives of the drug (whichever is longer). Traditional Chinese medicine with anti-tumor indications is within 2 weeks prior to the first dose of the study drug.
6. Patients who have received systemic corticosteroids (prednisone>10mg/day or equivalent doses of similar drugs) or other immunosuppressive treatments within 14 days prior to the first dose of the study drug; Excluding the use of local, ocular, intra-articular, intranasal, and inhaled corticosteroids for treatment; Short term use of corticosteroids for preventive treatment (such as preventing contrast agent allergies).
7. Taking live attenuated vaccines within 4 weeks prior to the first dose of the study drug, or it is expected that live attenuated vaccines will be vaccinated during the study period.
8. Participants who have previously received oncolytic virus therapy (such as T-vec, T3011, etc.), gene therapy, cell therapy, and tumor vaccines.
9. Participants have a history of splenectomy or organ transplantation.
10. Participants with the malignant tumors other than the disease treated in this study, except for the following:

    * Malignant tumors that have undergone treatment with the aim of cure, at least more than 5 years from the drug treatment, have no known active diseases, and have a low potential risk of recurrence;
    * Fully treated non-melanoma skin cancer or malignant freckle like nevi with no evidence of disease;
    * In situ cancer with sufficient treatment and no evidence of disease.
11. All toxicities caused by prior radiotherapy, chemotherapy or other treatments have recovered to Grade ≤1 (CTCAE 5.0) (except for alopecia), including but not limited to urinary tract infection, urinary tract irritation, and gross hematuria.
12. Indwelling ureteral stent or having a history of bladder ureteral reflux disease.
13. Major cardiovascular diseases, such as New York Heart Association heart disease (grade II or higher), myocardial infarction within the first three months of enrollment, unstable arrhythmia or unstable angina.
14. Having the history of autoimmune diseases, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wagner's granulomatosis, Sjogren's syndrome, Guillain Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. Except for patients with hypothyroidism or diabetes who have good control of alternative treatment.
15. Persistent or active infections exist, and drug treatment and control are still not ideal; Including but not limited to: active pulmonary tuberculosis, non negative AIDS virus (HIV) antibody, positive hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA) quantity ≥ the lower limit of the laboratory test in the research center, hepatitis C virus antibody (HCV Ab) positive and hepatitis C virus RNA quantity ≥ the lower limit of the laboratory test in the research center.
16. Participants who require oral or intravenous use of anti herpesvirus drugs during the study period (including but not limited to acyclovir, valaciclovir, penciclovir, famciclovir, ganciclovir, foxinkane, cedofovir, etc.) (excluding local use such as topical use).
17. Participants with the history of allergic reactions to HSV-1, IL-12, or anti PD-1 antibodies and similar biological components, or those known to have allergic reactions to any component of T3011.
18. Fever above 38.5 ℃ with no explained reason during the screening period, washout period/baseline period, or on the day of administration (the researcher determines that fever caused by tumors can be included), according to the researcher's judgment, may affect the patient's participation \in this trial or interfere with the evaluation of efficacy.
19. In the period of recurrent herpes simplex virus infection, there are corresponding clinical manifestations, such as lip herpes, herpetic keratitis, herpetic dermatitis, genital herpes, etc.
20. Participants who have previously developed non infectious pneumonia/interstitial pneumonia or are intolerant to immunotherapy drugs (including but not limited to anti PD-1/PD-L1 antibodies) (including but not limited to developing ≥ grade 3 immune related adverse events [irAEs]) (excluding endocrine related irAEs that can be stably controlled through hormone replacement therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
CR rate or relapse-free survival rates at 3, 6, 9 and 12 months after the first study dose | 3, 6, 9 and 12 months after first study dose
  Defined as the rate of Complete response or relapse-free survival at 3, 6, 9 and 12 months after first study drug administration
Recurrence-free survival, RFS | Up to 2 years
  Defined as relapse-free survival time
Progression-free survival, PFS | Up to 2 years
  Defined as time to progression-free survival
Incidence of radical cystectomy | Up to 2 years
  Defined as the rate at which radical cystectomy occurs
5-year survival rate | Up to 5 years
  Defined as survival rate at 5 year of administered treatment
Adverse Events, AE | up to 30 days after completion of treatment
  Evaluation standard is CTCAE V5.0
Serious Adverse Event, SAE | up to 30 days after completion of treatment
  Evaluation standard is CTCAE V5.0
Dose-limiting toxicity (DLT) events | First cycle of treatment, i.e. within 28 days of first instillation
  Defined as a toxic reaction related to the test drug occurring within the first cycle of treatment, i.e. within 28 days of the first instillation
Abnormal clinically significant vital signs and their incidence | Up to 1 years
  Abnormal clinically significant vital signs and their incidence
Abnormal clinically significant physical findings and their incidence | Up to 1 years
  Abnormal clinically significant physical findings and their incidence
Abnormal clinically significant laboratory findings and their incidence | Up to 1 years
  Abnormal clinically significant laboratory findings and their incidence

CONTACTS AND LOCATIONS:
Overall Officials: Dingwei Ye, Doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No